CLINICAL TRIAL: NCT06631469
Title: Behaviour-focused Personalised Nutrition Intervention to Promote Sustainable and Healthy Diets in University Students: a Feasibility Pilot Study
Brief Title: Behaviour-focused Personalised Nutrition Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: PLAN'EAT Consortium (https://planeat-project.eu/) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LS-23-72-Gibney; 101061023 (Other Grant/Funding Number: European Union Horizon Europe)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-10

CONDITIONS: Dietary Behaviours; Sustainable Healthy Diet; Personalised Nutrition
Keywords: Sustainable diet; Personalised nutrition; Dietary behaviours; University; Students

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Who Masked: Participant
Masking Description: Single-blinded parallel study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalised behavioural sustainable and healthy dietary recommendations (Experimental): Personalised dietary plan, standardised behavioural support (based on previous personalised nutrition trials and usual care in dietetic practice), plus personalised behavioural support and strategies aimed at meeting personalised dietary recommendations.
  Interventions: Behavioral: Personalised behavioural sustainable and healthy dietary recommendations
- Personalised sustainable and healthy dietary recommendations (Active Comparator): Personalised dietary plan and standardised behavioural support (based on previous personalised nutrition trials and usual care in dietetic practice) aimed at meeting personalised dietary recommendations.
  Interventions: Behavioral: Personalised sustainable and healthy dietary recommendations

INTERVENTIONS:
Behavioral: Personalised behavioural sustainable and healthy dietary recommendations — Personalised dietary plan and standardised behavioural support (based on previous personalised nutrition trials and usual care in dietetic practice), plus the addition of receiving personalised behavioural support and strategies.
  Arms: Personalised behavioural sustainable and healthy dietary recommendations
Behavioral: Personalised sustainable and healthy dietary recommendations — Personalised dietary plan and standardised behavioural support and strategies (based on previous personalised nutrition trials and usual care in dietetic practice).
  Arms: Personalised sustainable and healthy dietary recommendations

SUMMARY:
The aim of this study is to test the efficacy, feasibility, and acceptability of a novel, behaviour-focused personalised nutrition intervention compared to a control personalised nutrition intervention for improving adherence to sustainable and healthy dietary recommendations in university students.

DETAILED DESCRIPTION:
Participants will be recruited from the University College Dublin (UCD) PLAN'EAT Living Lab (LL) Citizen Panel which will form a separate registration. The UCD PLAN'EAT LL is a series of studies designed to develop, implement, and evaluate strategies to support University students' transition towards a sustainable healthy diet. The UCD PLAN'EAT LL study will recruit up to n=500 healthy students (aged 18-30 years) attending UCD, Belfield Campus, to join the UCD PLAN'EAT LL Citizen Panel. Upon successful screening and completion of informed consent, participants will be invited to join the UCD PLAN'EAT LL Citizen Panel and complete initial baseline data collection measures (which will be detailed in a separate registration). Following completion of this baseline data collection, participants within the UCD PLAN'EAT LL Citizen Panel will be subsequently invited to participate in this study detailed below.

Participants within the UCD PLAN'EAT LL Citizen Panel will be invited to participate in a 4-week study. This study will aim to recruit n=40 participants within the UCD PLAN'EAT LL Citizen Panel. After successful screening and informed consent, participants will be randomised into two separate groups (n=20 control group; n=20 intervention group) receiving different types of personalised recommendations and strategies using decision tree algorithms to support them to consume a healthier and more sustainable diet. The control group will receive a personalised dietary plan and standardised behavioural support (based on previous personalised nutrition trials and usual care in dietetic practice) to meet their personalised dietary recommendations. The intervention group will receive the same as the control group, with the addition of receiving personalised behavioural support and strategies to help them meet their personalised dietary recommendations.

Baseline: Participants will be asked to complete a questionnaire including questions on demographics, health, dietary behaviours, and lifestyle and a dietary assessment. The dietary assessment will include 3 online 24-hour dietary recalls (2 non-consecutive weekdays and 1 weekend day) (via the web-based dietary recall tool, Foodbook24).

Following completion of baseline measures, participants will be invited to attend a study visit in UCD. Participants will undergo a diet counselling session, where they will receive a personalised feedback report and advice from a nutritionist on how to achieve their goal of eating a more sustainable and healthy diet.

Midpoint: Participants will be contacted by a member of the research team via email or phone message to check their progression and to address any queries.

Endpoint: At the end of the 4-week study, participants will complete a diet-related questionnaire and a second dietary assessment. The dietary assessment will include 3 online 24-hour dietary recalls (2 non-consecutive weekdays and 1 weekend day) (via the web-based dietary recall tool, Foodbook24).

Following completion of endpoint measures, retention rates (number of participants who complete endpoint measures / number of participants enrolled into the study x 100) and data completion rates (number of complete datasets for each outcome measure / number of participants enrolled ×100) will be calculated to assess study feasibility and acceptability.

Process Evaluation:

At the end of this study, all participants will be invited to complete a study evaluation questionnaire including feasibility, acceptability, and engagement measures. In addition, a subsample of participants will also be invited to participate in focus groups or one-to-one interviews to explore topics on study feasibility encompassing, for example, their study experience, study acceptability, factors affecting participation rates (e.g., barriers/ enablers), study engagement, and suggestions for improvement. The focus groups or one-to-one interviews will be guided by the APEASE (Acceptability, Practicality, Effectiveness, Affordability, Side-effects, Equity) criteria.

ELIGIBILITY:
Student Participants:

Inclusion Criteria:

* Be a UCD student (aged 18-30 years) attending Belfield Campus.
* Be an adult between the age of 18-30 years old, and in general good health.

Exclusion Criteria:

* Do not attend UCD Belfield Campus.
* Are under 18 years of age or over 30 years of age.
* Have a diagnosis of an acute or chronic medical condition that could interfere with the outcomes of the study. Such diagnosis include (but not limited to) cardiovascular disease, diabetes mellitus, cancers (within the past 5 years), etc.
* Are pregnant, lactating or planning to become pregnant.
* Are following a medically prescribed diet.
* Are immunocompromised or have a suspected immunodeficiency.
* Have a known food allergy.
* Taking part in another diet-related research study that could interfere with the outcomes of this study
* Consume ≥2 servings per day of legumes.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Legume intake (grams per day) | 4 weeks
  Participants will record their diet at baseline (habitual diet) and endpoint (intervention diet) using an online 24-hour recall method. Legume intake will be calculated using dietary intake records (baseline: 3x 24-hour recalls; endpoint: 3x 24-hour recalls). The primary outcome measure is the change in legume intake (g/ day) as a result of the intervention diet.

SECONDARY OUTCOMES:
Plant-based food intake (grams per day) | 4 weeks
  Participants will record their diet at baseline (habitual diet) and endpoint (intervention diet) using an online 24-hour recall method. Plant-based food intake will be calculated using dietary intake records (baseline: 3x 24-hour recalls; endpoint: 3x 24-hour recalls). The secondary outcome measure is the change in plant-based food intake (g/ day) as a result of the intervention diet.
Fruit intake (grams per day) | 4 weeks
  Participants will record their diet at baseline (habitual diet) and endpoint (intervention diet) using an online 24-hour recall method. Fruit intake will be calculated using dietary intake records (baseline: 3x 24-hour recalls; endpoint: 3x 24-hour recalls). The secondary outcome measure is the change in fruit intake (g/ day) as a result of the intervention diet.
Vegetable intake (grams per day) | 4 weeks
  Participants will record their diet at baseline (habitual diet) and endpoint (intervention diet) using an online 24-hour recall method. Vegetable intake will be calculated using dietary intake records (baseline: 3x 24-hour recalls; endpoint: 3x 24-hour recalls). The secondary outcome measure is the change in vegetable intake (g/ day) as a result of the intervention diet.
Meat intake (grams per day) | 4 weeks
  Participants will record their diet at baseline (habitual diet) and endpoint (intervention diet) using an online 24-hour recall method. Meat intake will be calculated using dietary intake records (baseline: 3x 24-hour recalls; endpoint: 3x 24-hour recalls). The secondary outcome measure is the change in meat intake (g/ day) as a result of the intervention diet.
High fat, sugar, salt (HFSS) food intake (grams per day) | 4 weeks
  Participants will record their diet at baseline (habitual diet) and endpoint (intervention diet) using an online 24-hour recall method. High fat, sugar, and salt food intake will be calculated using dietary intake records (baseline: 3x 24-hour recalls; endpoint: 3x 24-hour recalls). The secondary outcome measure is the change in high fat, sugar, and salt food intake (g/ day) as a result of the intervention diet.

OTHER OUTCOMES:
Feasibility | 4 weeks
  Following completion of endpoint measures, retention rates (number of participants who complete endpoint measures / number of participants enrolled into the study x 100) will be calculated to assess study feasibility and acceptability.
Feasibility | 4 weeks
  Following completion of endpoint measures, data completion rates (number of complete datasets for each outcome measure / number of participants enrolled × 100) will be calculated to assess study feasibility and acceptability.
Diet-related greenhouse gas emissions reported as kilograms of carbon dioxide equivalents per day | 4 weeks
  Participants will record their diet at baseline (habitual diet) and endpoint (intervention diet) using an online 24-hour recall method. Diet-related greenhouse gas emissions will be estimated using food, nutrient and food-related greenhouse gas emission databases (measured as kilograms of carbon dioxide equivalents). The tertiary outcome measure is the change in diet-related greenhouse gas emissions (kgCO2-eq/day) as a result of the intervention diet.
Self-reported behavioural automaticity index | 4 weeks
  Participants will record their self-reported behavioural automaticity at baseline and endpoint via a questionnaire. Each participant's score can range from 4-28 (with 4 indicating low behavioural automaticity and 28 indicating high behavioural automaticity). The quaternary outcome measure is the change in participants self-reported behavioural automaticity as a result of the intervention.
Process Evaluation | 4 weeks
  At the end of this study, participants will complete an evaluation questionnaire. A subsample of participants will be invited to participate in focus groups or one-to-one interviews. Participants will evaluate study feasibility on topics encompassing: study experience, study acceptability, factors affecting participation rates (barriers and enablers), study engagement and suggestions for improvement. The quinary outcome is participants evaluation of this study.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
At the beginning of the study, each participant will have a study code assigned to them. All data collected from the study will be stored using these unique study codes. A file will be set up which will be stored in a separate location to the study data. This file will contain a list which will link each participants contact details to the corresponding ID code. All stored information will be password-protected and only accessible to the research team/ named researchers on the project. Pseudonymised/ anonymised data will be shared with PLAN'EAT partners where appropriate.

REFERENCES:
- [Background] Davies KP, Gibney ER, Leonard UM, Lindberg L, Woodside JV, Kiely ME, Nugent AP, Arranz E, Conway MC, McCarthy SN, O'Sullivan AM. Developing and testing personalised nutrition feedback for more sustainable healthy diets: the MyPlanetDiet randomised controlled trial protocol. Eur J Nutr. 2024 Oct;63(7):2681-2696. doi: 10.1007/s00394-024-03457-0. Epub 2024 Jul 6. PMID 38970665
- [Background] Macready AL, Fallaize R, Butler LT, Ellis JA, Kuznesof S, Frewer LJ, Celis-Morales C, Livingstone KM, Araujo-Soares V, Fischer AR, Stewart-Knox BJ, Mathers JC, Lovegrove JA. Application of Behavior Change Techniques in a Personalized Nutrition Electronic Health Intervention Study: Protocol for the Web-Based Food4Me Randomized Controlled Trial. JMIR Res Protoc. 2018 Apr 9;7(4):e87. doi: 10.2196/resprot.8703. PMID 29631993
- [Background] Writing Group of the Nutrition Care Process/Standardized Language Committee. Nutrition care process and model part I: the 2008 update. J Am Diet Assoc. 2008 Jul;108(7):1113-7. doi: 10.1016/j.jada.2008.04.027. No abstract available. PMID 18589014
- [Background] Rigby RR, Mitchell LJ, Hamilton K, Williams LT. The Use of Behavior Change Theories in Dietetics Practice in Primary Health Care: A Systematic Review of Randomized Controlled Trials. J Acad Nutr Diet. 2020 Jul;120(7):1172-1197. doi: 10.1016/j.jand.2020.03.019. Epub 2020 May 20. PMID 32444328
- See also: British Dietetic Association. Model and Process for Nutrition and Dietetic Practice. British Dietetic Association; 2021. — https://www.bda.uk.com/practice-and-education/nutrition-and-dietetic-practice/professional-guidance/model-and-process-for-dietetic-practice.html
- See also: Michie S, Atkins L, West R. The Behaviour Change Wheel: A Guide to Designing Interventions. Great Britain: Silverback Publishing; 2014. — https://www.behaviourchangewheel.com/